CLINICAL TRIAL: NCT03140267
Title: Assessment of the Evolution of Force and Endurance of Inspiratory Muscles in Intubated and Mechanically-ventilated ICU Patients With Difficult Weaning
Brief Title: Assessment of Inspiratory Muscles Strength and Endurance Evolution on Difficult to Wean Patients in Intensive Care Unit
Acronym: EFES
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CHUBX 2015/37
Record Dates: First submitted 2017-05-02; First posted 2017-05-04 (Actual); Last update posted 2020-05-13 (Actual); Status verified 2020-05

CONDITIONS: Weaning From Mechanical Ventilation
Keywords: Ventilated induced diaphragmatic dysfunction; Weaning; Inspiratory muscle training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Difficult to wean patients (Experimental): Maximal Inspiratory Pressure and Peak Pressure from the inclusion day to the extubation day will be measure.
  Interventions: Diagnostic Test: Difficult to wean patients

INTERVENTIONS:
Diagnostic Test: Difficult to wean patients — Subjects will be following during 18 hours in an invasive mechanical ventilation in a controlled mode. After failure of first single breath trial during 2 hours and presence of sevrability criterias defined by the European consensus conference in 2007, Maximal Inspiratory Pressure and Peak Pressure will be measure.

SUMMARY:
Ventilator-induced diaphragmatic dysfunction appears to contribute to slow weaning from mechanical ventilation. Several trials of inspiratory muscle training to facilitate weaning in intensive care have been performed, with inconsistent results, utilizing different methods of IMT in different populations.

To perform the best IMT program, we need to know the physio-pathology of the diaphragm in difficult to wean patients.

This study proposes to discriminate the two main characteristics of the inspiratory muscles: strength and endurance.

By analyzing the evolution of strength and endurance during all the weaning period, we want to know which characteristic has the more deficiency to adapt in a second time an effective program of IMT.

DETAILED DESCRIPTION:
The main objective of this study is to determinate which characteristic of inspiratory muscles between strength and endurance has more deficiency in difficult to wean patients. In a second time, the results of this study will help to choose the best IMT program to assess his impact on the weaning time.

We are going to conduct an interventional trial because of Peak Pressure measure, which is not measure in care practice. Following 18h of invasive mechanical ventilation in a controlled mode, the failure of the first single breathe trial of 2 hours and the presence of sevrability criterias defined by the European consensus conference in 2007, 80 participants will be included in the medical intensive care unit of Bordeaux's hospital. We'll perform measurements of the Maximal Inspiratory Pressure and Peak Pressure from the inclusion to the extubation.

ELIGIBILITY:
Inclusion Criteria:

* Patient ventilated more than 18h in a controlled mode;
* First single breathe trial of 2 hours failure;
* Presence of sevrability criterias definied by the European consensus conference in 2007 as usually used:

  * diminution of the sedfative agents ;
  * Patients with spontaneous beath in VAC mode or patient ventilated in a VSAI-PEP mode;
  * PaO2/FiO2 ≥150;
  * Absence d'inotropes ou de vasopresseurs à forte dose ou dose croissante (<1mg/h);
  * SaO2 > 90% with FiO2 ≤ 50%;
  * PEP ≤ 8cmH2O;
  * Corporal température between 36°C and 39°C;
  * Glasgow Score ≥ 8;
* Patient or family consent.

Exclusion Criteria:

* Age < 18 years ;
* medically unstable;
* Poor vital pronostic at very short term;
* Cardiac arrest with a poor neurological prognostic;
* Neuromuscular disease ;
* Tracheostomy ;
* Current pregnancy ;
* Patients with guardianship or trusteeship.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2017-05-14 (Actual); Primary Completion 2020-01-23 (Actual); Study Completion 2020-01-23 (Actual)

PRIMARY OUTCOMES:
Maximal Inspiratory Pressure score assessment | Daily measure (from inclusion day (day 1) to extubation day (maximum day 28))
  Correlation between Maximal Inspiratory Pressure score assessment (inspiratory muscle strength index) and duration of weaning period

SECONDARY OUTCOMES:
Peak Pressure assessment | Each 7 days (from inclusion day (day 1) to extubation day (maximum day 28))
  Correlation between Peak Pressure assessment (inspiratory muscle endurance index) and duration of weaning period
Maximal Inspiratory Pressure score assessment after weaning success | From inclusion day (day 1) to extubation success day (maximum day 28)
  Correlation between Maximal Inspiratory Pressure score assessment and weaning success (not re-intubated in the 48h post-extubation)
Peak Pressure assessment after weaning success | From inclusion day (day 1) to extubation success day (maximum day 28)
  Correlation between Peak Pressure assessment and weaning success.
Maximal Inspiratory Pressure score assessment and hospitalization | From inclusion day (day 1) to come out of hospital day (maximum day 30)
  Correlation between Maximal Inspiratory Pressure score assessment and intensive care unit length
Peak Pressure assessment and hospitalization | From inclusion day (day 1) to come out of hospital day (maximum day 30)
  Correlation between Peak Pressure assessment and intensive care unit length
Adverses events | Daily measures (from inclusion day (day 1) to come out of hospital day (maximum day 30))
  Adverses events occur during Maximal Inspiratory Pressure and Peak Pressure measures

CONTACTS AND LOCATIONS:
Overall Officials: Perez Paul, Dr, Study Chair — USMR
Locations (2):
- France (2):
  - Hôpital Haut-Lévêque, Bordeaux
  - Hôpital Pellegrin, Bordeaux

IPD SHARING:
Plan to Share IPD: No